CLINICAL TRIAL: NCT05752305
Title: Effect of Preoperative Administration of Dexamethasone Versus Methylprednisolone in Surgical Extraction of Retained Lower Third Molars
Brief Title: Use of Corticosteroids in Third Molar Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Unai Fernández Martín, Principal Investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3180/CEIH/2023
Record Dates: First submitted 2023-02-09; First posted 2023-03-02 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Inflammation; Pain, Postoperative; Trismus
MeSH Terms: conditions — Inflammation; Pain, Postoperative; Trismus | interventions — Dexamethasone; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methylprednisolone group (Experimental): Preoperative administration of 40mg of methylprednisolone via submucosa
  Interventions: Drug: MethylPREDNISolone 40 Mg/mL Injectable Suspension
- Dexamethasone group (Experimental): Preoperative administration of 8mg of dexamethasone via submucosa
  Interventions: Drug: Dexamethasone 4 Mg/mL Injectable Solution

INTERVENTIONS:
Drug: Dexamethasone 4 Mg/mL Injectable Solution — Preoperative submucosal administration of 8mg of dexamethasone or 40mg of methylprednisolone.
  Arms: Dexamethasone group
Drug: MethylPREDNISolone 40 Mg/mL Injectable Suspension — Preoperative submucosal administration of 8mg of dexamethasone or 40mg of methylprednisolone.
  Arms: Methylprednisolone group

SUMMARY:
Surgical extraction of retained lower third molars is associated with the development of postoperative complications, including inflammation, trismus and postoperative pain, that lead to a decrease in patients' quality of life. Therefore, the use of drugs is essential to reduce the morbidity associated with surgery, with NSAIDs and corticosteroids being the most commonly used drugs.

DETAILED DESCRIPTION:
Surgical extraction of retained lower third molars is associated with the development of postoperative complications, including inflammation, trismus and postoperative pain. Traditionally, NSAIDs have been used for the treatment of postoperative pain and inflammation, although corticosteroids are increasingly used in oral surgery, as they have proven to be clinically effective in reducing postoperative complications without causing serious adverse effects. Although numerous studies have been carried out comparing different corticosteroids in order to determine which of them is the most effective, there is still no clinical protocol regulating the use of these drugs in oral surgery. Therefore, this clinical trial is based on comparing two of the most studied corticosteroids used in oral surgery to date: dexamethasone and methylprednisolone.

This study is based on the preoperative administration of 8mg of dexamethasone or 40mg of methylprednisolone via submucosa, randomly, in patients undergoing surgical extraction of a retained lower third molar, to determine which of these two drugs is more effective in the prevention of inflammation, trismus and postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Indication for surgical extraction of a retained lower third molar

Exclusion Criteria:

* Patients treated with corticosteroids in the last 3 months
* Patients treated with NSAIDs in the last 7 days
* Patients with hypersensitivity to the drug
* Patients with a medical condition that contraindicates the administration of the drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-01-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Postoperative inflammation following third molar surgical extraction | 7 days
  Postoperative swelling was determined by measuring tragus-chin distance, tragus-labial cleft distance and eye angle-jaw angle distance, using a millimeter ruler.
Postoperative trismus following third molar surgical extraction | 7 days
  Postoperative trismus was assessed by measuring the patient's maximum mouth opening (measuring the distance between the incisal edge of the upper central incisor and the lower central incisor) using a millimeter ruler.
Postoperative pain following third molar surgical extraction | 7 days
  Postoperative pain was measured using the Visual Analogue Scale (VAS): patients were asked to assign a numerical value from 0-100 (0 being no pain and 100 the maximum pain).

CONTACTS AND LOCATIONS:
Overall Officials: Unai Fernández, Principal Investigator — Universidad de Granada
Locations (1):
- Unai Fernández Martín, Granada, Spain

IPD SHARING:
Plan to Share IPD: No